CLINICAL TRIAL: NCT00002109
Title: Double-Blind Study of Timunox (Thymopentin) in Asymptomatic HIV-Infected Patients Receiving Either Mono (AZT or ddI) or Combination (AZT/ddI or AZT/ddC) Anti-Retroviral Therapy
Brief Title: Double-Blind Study of Timunox (Thymopentin) in Asymptomatic HIV-Infected Patients Receiving Either Mono (AZT or ddI) or Combination (AZT / ddI or AZT / ddC) Anti-Retroviral Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Immunobiology Research Institute (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 015H; 07.32.033-93
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: HIV Infections
Keywords: Thymopentin; Zalcitabine; Didanosine; Drug Therapy, Combination; Zidovudine; Stavudine
MeSH Terms: conditions — HIV Infections | interventions — Thymopentin; Stavudine; Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Thymopentin
Drug: Stavudine
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To confirm results from a previous study in which the combination of thymopentin plus zidovudine ( AZT ), an antiretroviral agent, slowed disease progression in HIV-infected asymptomatic patients. To evaluate the efficacy and safety of thymopentin in HIV-infected asymptomatic patients receiving either monotherapy with AZT, didanosine ( ddI ), or stavudine ( d4T ), or combination antiretroviral therapy with AZT / ddI or AZT / zalcitabine ( ddC ).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Asymptomatic HIV infection.
* CD4 count 100-400 cells/mm3.
* No HIV-associated neurologic abnormalities or constitutional symptoms.
* No oral hairy leukoplakia.
* At least 6 months of prior AZT.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Abnormal chest x-ray, consistent with active opportunistic infection.
* Hypersensitivity to thymopentin.
* Significant chronic underlying medical illness.
* Grade 2 or worse peripheral neuropathy.

Concurrent Medication:

Excluded:

* HIV vaccines.
* Investigational or non-FDA approved medication.
* Immunomodulatory therapies.
* Experimental therapies.
* Any antiretroviral therapy other than AZT, ddI, ddC, d4T, or 3TC.

Patients with the following prior conditions are excluded:

* Herpes zoster (within the past year).
* Recurrent (> one episode) oral candidiasis (confirmed).
* Vulvovaginal candidiasis (persistent, frequent, or poorly responsive to therapy).
* Bacillary angiomatosis.
* Listeriosis.
* Idiopathic thrombocytopenia purpura.

Prior Medication:

Excluded at any time prior to study entry:

More than one dose of thymopentin.

Excluded within 30 days prior to study entry:

* HIV vaccines.
* Investigational or non-FDA approved medication.
* Immunomodulatory therapies.
* Experimental therapies.
* Any antiretroviral therapy other than AZT, ddI, ddC, d4T, or 3TC.

Required:

* Prior AZT (>= 300 mg/day) for at least 6 months; on current regimen (any combination of approved nucleoside analogues) for at least 4 weeks.

Significant active alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (50):
- United States (48):
  - Fisher Med Group, Phoenix, Arizona
  - Ctr for Special Immunology, Irvine, California
  - Beer Med Group, Los Angeles, California
  - Gottlieb Med Group, Pasadena, California
  - AIDS Community Research Consortium, Redwood City, California
  - HIV Research Group, San Diego, California
  - Conant Med Group, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Pacific Oaks Med Group, Sherman Oaks, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Dr Gary Blick, Greenwich, Connecticut
  - Dr Larry Bruni, Washington D.C., District of Columbia
  - Novum Inc, Washington D.C., District of Columbia
  - Community Research Initiative, Coral Gables, Florida
  - Ctr for Special Immunology, Fort Lauderdale, Florida
  - Stratogen of Ft Lauderdale, Fort Lauderdale, Florida
  - Stratogen of South Florida, Miami Beach, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Saint Joseph's Hosp / Infectious Disease Rsch Institute, Tampa, Florida
  - West Paces Clinical Research Inc, Atlanta, Georgia
  - Northwestern Univ Med Ctr, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Ctr for Special Immunology, Chicago, Illinois
  - Infectious Diseases Research Clinic / Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - CRI of New England, Brookline, Massachusetts
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Systemic Mycoses Pathogen Study Group / Wash Univ Sch of Med, St Louis, Missouri
  - Lovelace Scientific Resource, Albuquerque, New Mexico
  - Dr David DiPietro, New York, New York
  - Ctr for Special Immunology, New York, New York
  - Dr Howard A Grossman, New York, New York
  - Dr Patrick Hennessey, New York, New York
  - New York Hosp - Cornell Med Ctr, New York, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Van Etten Hosp / Bronx Municipal Hosp Ctr, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Associates Med and Mental Health, Tulsa, Oklahoma
  - Dr Joel Godbey, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Graduate Hosp, Philadelphia, Pennsylvania
  - Novum Inc, Pittsburgh, Pennsylvania
  - Central Texas Med Foundation, Austin, Texas
  - Dr Christopher McNulty, Dallas, Texas
  - Nelson-Tebedo Community Clinic, Dallas, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Novum Inc, Kirkland, Washington
- Puerto Rico (2):
  - Univ of Puerto Rico Med Sciences Campus, Rio Piedras
  - Initiativa Comunitaria de Investigacion, San Juan